CLINICAL TRIAL: NCT00972712
Title: A Phase I Protocol of the Combination Bortezomib and Tipifarnib for Relapsed or Refractory Multiple Myeloma
Brief Title: Protocol of the Combination of Bortezomib and Tipifarnib for Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Ortho Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Sagar Lonial, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000655; WCI1192-06 (Other: Other)
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Bortezomib and Tipifarnib
  Interventions: Drug: Bortezomib and Tipifarnib

INTERVENTIONS:
Drug: Bortezomib and Tipifarnib — Dose level -1: Bortezomib (0.7 mg/m²; days 1,4,8,11); Tipifarnib (100 mg po BID)
  Dose level 1: Bortezomib (1.0 mg/m²; days 1,4,8,11); Tipifarnib (100 mg po BID)
  Dose level 2: Bortezomib (1.0 mg/m²; days 1,4,8,11); Tipifarnib (200 mg po BID)
  Dose level 3: Bortezomib (1.0 mg/m²; days 1,4,8,11); Tipifarnib (300 mg po BID)
  Dose level 4: Bortezomib (1.0 mg/m²; days 1,4,8,11); Tipifarnib (400 mg po BID)
  Schema B
  Dose level 1: Bortezomib (1.3 mg/m²; Days 1,4,8,11); Tipifarnib (300 mg po BID)
  Dose level 2: Bortezomib (1.3 mg/m²; Days 1,4,8,11); Tipifarnib (400 mg po BID)
  Other Names: Velcade; Zarnestra

SUMMARY:
The purpose of this study is to test the effect of the combination of bortezomib and tipifarnib. Bortezomib (VELCADE) is approved by the Food and Drug Administration (FDA) for the treatment of multiple myeloma patients who have received at least one prior therapy. Tipifarnib is not yet approved by the FDA and is an investigational drug. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. Because these drugs have not been used together before, it is not clear which dose of each agent is optimal when used in combination.

This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational drug. Phase I studies also try to define the appropriate dose of the investigational drugs to use for further studies. The investigators will test the safety of BORTEZOMIB and TIPIFARNIB together and see what effects (good and bad) it has on you and your MULTIPLE MYELOMA, and to find the highest dose of both agents that can be given without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study must meet criteria for relapsed or refractory multiple myeloma. Relapsed myeloma is defined in patients as increasing M-Spike or plasmacytoma compared to a previous measurement confirmed on at least two different settings. Refractory myeloma is defined as progression of disease on current therapy, and having received at least two courses of treatment with or without the use of high dose therapy and autologous transplant.
* Patients must have received at least 2 prior lines of therapy in order to be eligible for this treatment.
* Must be ≥ 18 years of age. Because no dosing or adverse event data are currently available on the use of bortezomib in combination with tipifarnib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric phase 1 combination trials.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2 (Karnofsky ≥ 60%, see Appendix A).
* Life expectancy of greater than 12 weeks.
* Patients must have organ and marrow function as defined below:

  * Leukocytes ≥ 1,000/microliter (mcL)
  * Absolute neutrophil count ≥ 500/mcL
  * Platelets ≥ 25,000/mcL
  * Total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine ≤ 2.5 OR
  * Creatinine clearance ≥ 20 mL/min/1.73 m² for patients with creatinine levels above institutional normal.
* Eligibility of patients receiving any medications or substances with the potential or known to affect the activity or pharmacokinetics of bortezomib or tipifarnib will be determined following review of their case by the Principal Investigator. Patients must be on bisphosphonates therapy unless precluded by osteonecrosis of the jaw (ONJ) or other clinical circumstances at the investigators discretion. Patients may receive erythroid growth factors as needed, per institutional guidelines. Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs) (e.g., phenytoin, carbamazepine, phenobarbital) nor any other cytochrome P450 3A4 (CYP3A4) inducer such as rifampin or St. John's wort.
* The effects of bortezomib and tipifarnib on the developing human fetus are unknown. For this reason, women with child-bearing potential and men must agree to use adequate contraception prior to entering the study. Adequate contraception includes hormonal therapy, a barrier method of birth control or abstinence. Appropriate contraception must be used for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately, and will be immediately discontinued from the study. Any woman who becomes pregnant during the study will be followed throughout their pregnancy until its outcome (i.e. delivery, still birth, miscarriage).

  * Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
  * Male subject agrees to use an acceptable method of contraception for the duration of the study.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to boronic acid, bortezomib, tipifarnib, or other agents used in study. Known allergy to imidazole drugs, such as clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, isoconazole, sulconazole, tioconazole or terconazole.
* Patients with a poorly controlled intercurrent illness will be excluded including but not limited to those with ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social climate that would limit compliance with study requirements.
* Pregnant women are excluded from this study because bortezomib and tipifarnib are Class D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bortezomib and tipifarnib, breastfeeding should be discontinued if the mother is treated with bortezomib and tipifarnib. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with bortezomib and tipifarnib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Other Exclusion Criteria

* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment.
* Patient has hypersensitivity to boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum ß-human chorionic gonadotropin (ß-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Adverse events based on the NCI Common Terminology Criteria (CTC) version 3.0 | Ongoing from start of treatment until 30 days post

SECONDARY OUTCOMES:
Laboratory tests to include: serum protein electrophoresis, quantitative immunoglobulins assay and immunofixation, 24 hour urine collection for Bence Jones protein, total proteins, and creatinine, bone marrow aspiration and analysis for plasma cells | Every 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Lonial, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (2):
  - City of Hope Cancer Institute, Duarte, California
  - Emory University Winship Cancer Institute, Atlanta, Georgia
- Princess Margaret Cancer Center, Toronto, Ontario, Canada